CLINICAL TRIAL: NCT01992822
Title: Experimental Pain Sensitivity of Subjects With Fibromyalgia Before and After rTMS Treatment in Relation to the Clinical Improvement
Brief Title: Pain Sensitivity of Subjects With Fibromyalgia Before and After Repetitive Transcranial Magnetic Stimulation Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Esquirol (Other)
Responsible Party: Principal Investigator, Dominique Malauzat, MD, Centre Hospitalier Esquirol
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2013-A01508-37
Record Dates: First submitted 2013-11-19; First posted 2013-11-25 (Estimated); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Fibromyalgia
Keywords: rTMS; fibromyalgia; experimental pain
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- experimental pain induction (Experimental): application of a pre-fixed pressure (160 kPa) on the forearm
  Interventions: Other: experimental pain induction

INTERVENTIONS:
Other: experimental pain induction — application of a pre-fixed pressure (160 kPa) on the forearm.

SUMMARY:
The principal study aims at evaluating the efficiency of rTMS maintenance sessions on the clinical effect of a rTMS cure in fibromyalgic subjects. This complementary study consists in the evaluation of the experimental sensitivity to mechanical pain (pressure application on the forearm) of subjects presenting fibromyalgia before and after rTMS treatment (21 days), and to put the results in relation to the clinical improvement and the psychometric evaluations (depression,fibromyalgia impact questionnaire, catastrophism).

ELIGIBILITY:
* Inclusion Criteria:

presence of the criteria from the American College of Rheumatology (2010)for fibromyalgia diagnosis, painful state for more than six months, visual analogic scale evaluation > or = 5, age between 18 and 70, no modification in therapeutic treatment one month before and during the protocol presence of actual or prior antalgic chronic treatment : pregabalin, duloxetine, milnacipran, gabapentin, venlafaxine, laroxyl, grade 1 or 2 antalgic residence in Limoges or the periphery, or the ability to come to the hospital for the treatment

Exclusion Criteria:

presence of non stabilized psychiatric comorbidity (personality trouble, addiction, suicide attempt, non controlled affective trouble), active epilepsy, previous cerebral traumatism, or cerebral surgery, intra-cranial hyper tension, pacemaker, metallic pieces in the brain, cochlear ocular implant, or any metallic material contra indicating magnetic resonance imaging.

clozapine, bupropion, methadon, theophyllin, or other non chemical antalgic technic established during the previous month(kinesitherapy, relaxation, hypnosis...), pregnancy, or administrative and judiciary protection, absence of health insurance.

known latex allergy, peripheral neuropathy, nerve lesion or dermatosis at the upper extremities, muscular lesion or pathology at the upper members, use of illicit drugs 48 hours before experimental pain test, use of antalgic or analgesic drug aiming at a punctual treatment during the prior 24 hours.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2013-11; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Variation in the Visual Analogic Scale (VAS)score after fixe pressure application (160 kPa) between the first rTMS session (T0) and the last rTMS session (T21)in relation to clinical improvement | 21 days
  The clinical improvement is defined as :
  30% decrease in the general painful state evaluated by VAS between T0 and T21 and response to the Patient's Global Impression of Change ≥ 6 at T21

SECONDARY OUTCOMES:
variation in the experimental pain feeling (VAS) between T0 and T21 in relation to treatment group | 21 days
variation in experimental pain feeling between T0 and T210 (the end of rTMS maintenance sessions) | 210 days
variation in Beck Depression Inventory scores between T0 and T21 | 21 days
variation in Fibromyalgia Impact Questionnaire score between T0 and T21 | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Malauzat, MD, Principal Investigator — CH Esquirol
Locations (1):
- Centre Hospitalier esquirol, Limoges, France